CLINICAL TRIAL: NCT00654316
Title: A Phase I Study of the Safety and Immunogenicity of BCG (Bacille Calmette-Guerin) Vaccine Delivered Intradermally by a Needle Injection in Healthy Volunteers Who Have Previously Received BCG.
Brief Title: Study of the Safety and Immunogenicity of Bacille Calmette Guerin (BCG) Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Dr Helen McShane, University of Oxford
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TB006
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-03

CONDITIONS: TB
Keywords: TB; Tuberculosis; MVA85A; Vaccine; BCG
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): BCG delivered intradermally into the deltoid region in volunteers who have received BCG 10 - 20 years previously.
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: BCG — intradermal injection of 0.1ml BCG over the deltoid muscle
  Other Names: Bacille Calmette-Guerin

SUMMARY:
Tuberculosis (TB) kills about three million people annually. It is estimated that one third of the world's population are latently infected with Mycobacterium tuberculosis (M.tb). Multi-drug resistant strains of M.tb, and co-infection with M.tb and HIV present major new challenges. The currently available vaccine, M. bovis BCG, is largely ineffective at protecting against adult pulmonary disease in endemic areas and it is widely agreed that a new more effective tuberculosis vaccine is a major global public health priority1. However, it may be unethical and impractical to test and deploy a vaccine strategy that does not include BCG, as BCG does confer worthwhile protection against TB meningitis and leprosy. An immunisation strategy that includes BCG is also attractive because the populations in which this vaccine candidate will need to be tested will already have been immunised with BCG.

M.tb is an intracellular organism. CD4+ Th1-type cellular responses are essential for protection and there is increasing evidence from animal and human studies that CD8+ T cells also play a protective role2. However, it has generally been difficult to induce strong cellular immune responses in humans using subunit vaccines. DNA vaccines induce both CD4+ and CD8+ T cells and thus offer a potential new approach to a TB vaccine. DNA vaccines encoding various antigens from M. tuberculosis have been evaluated in the murine model, and to date no DNA vaccine alone has been shown to be superior to BCG.

A heterologous prime-boost immunisation strategy involves giving two different vaccines, each encoding the same antigen, several weeks apart. Such regimes are extremely effective at inducing a cellular immune response. Using a DNA- prime/MVA-boost immunisation strategy induces high levels of CD8+ T cells in animal models of malaria and HIV5, and high levels of both CD4+ and CD8+ T cells in animal models of TB. BCG immunisation alone induces only CD4+ T cells in mice. A prime-boost strategy using BCG as the prime and a recombinant MVA encoding an antigen from M.tb that is also present in BCG (antigen 85A: 'MVA85A') as the boost, induces much higher levels of CD4+ T cells than BCG or MVA85A alone. In addition, this regime generates specific CD8+ T cells that are undetectable following immunisation with BCG alone.

DETAILED DESCRIPTION:
Recombinant viruses as vaccines.

Recombinant viruses used alone have for some years represented a promising vaccine delivery system, particularly for inducing cellular immune responses8. The recombinant virus encodes the immunising protein or peptide. Immunisation by a recombinant virus vaccine occurs when host cells take up and express the inoculated attenuated virus encoding a protective antigen. The expressed protein often has the native conformation, glycosylation, and other post-translational modifications that occur during natural infection. Recombinant viral vaccines may elicit both antibody and cytotoxic T-lymphocyte responses, which persist without further immunisations.

Many viruses have been investigated as potential recombinant vaccines. The successful worldwide eradication of smallpox via vaccination with live vaccinia virus highlighted vaccinia as a candidate for recombinant use. The recognition in recent years that non-replicating strains of poxvirus such as MVA and avipox vectors can be more immunogenic than traditional replicating vaccinia strains has enhanced the attractiveness of this approach. MVA (modified vaccinia virus Ankara) is a strain of vaccinia virus which has been passaged more than 570 times though avian cells, is replication incompetent in human cell lines and has a good safety record. It has been administered to more than 120,000 vaccinees as part of the smallpox eradication programme, with no adverse effects, despite the deliberate vaccination of high risk groups. This safety in man is consistent with the avirulence of MVA in animal models. MVA has six major genomic deletions compared to the parental genome severely compromising its ability to replicate in mammalian cells. Viral replication is blocked late during infection of cells but importantly viral and recombinant protein synthesis is unimpaired even during this abortive infection. Replication-deficient recombinant MVA has been seen as an exceptionally safe viral vector. When tested in animal model studies recombinant MVAs have been shown to be avirulent, yet protectively immunogenic as vaccines against viral diseases and cancer. The most useful data on the safety and efficacy of various doses of a recombinant MVA vaccine comes from clinical trial data with a recombinant MVA expressing a number of CTL epitopes from Plasmodium falciparum pre-erythrocytic antigens fused to a complete pre-erythrocytic stage antigen, Thrombospondin Related Adhesion Protein (TRAP). These trials have given a total of 169 immunisations with this recombinant MVA, to 49 UK vaccinees 38 Gambian vaccines (20 of whom were children aged 1-5). 6 doses of 1 x 10^7 pfu, 139 doses of 5 x 10^7 pfu, 6 doses of 1 x 10^8 pfu and 18 doses of 2.5 x 10^8 pfu have been administered, all without serious adverse effects.

Recombinant MVA encoding antigen 85A

Secreted antigens from M. tuberculosis are released from actively metabolising bacteria, and are important targets in protective immunity. Antigen 85A is a major secreted antigen from M. tuberculosis which forms part of the antigen 85 complex (A, B and C). This complex constitutes a major portion of the secreted proteins of both M.tb and BCG. It is involved in fibronectin binding within the cell wall and has mycolyltransferase activity.

MVA85A induces both a CD4+ and a CD8+ epitope when used to immunise mice. When mice are primed with BCG and then given MVA85A as a boost, the levels of CD4+ and CD8+ T cells induced are higher than with either BCG or MVA85A alone.

We are evaluating the safety and immunogenicity of the following 3 groups:

1. BCG alone
2. MVA85A alone
3. BCG prime-MVA85A boost

BCG-BCG provides a control group for BCG-MVA85A. Many countries have a tradition of repeated BCG vaccination and the criteria for revaccination differ between countries.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18-55 years.
* Normal medical history and physical examination.
* Normal urine dipstick, blood count, liver enzymes, and creatinine.

Exclusion Criteria:

* Exposure to TB at any point. A positive ESAT6/CFP10 Elispot response (defined as greater than 5 spots/well above background and at least double the background response).
* Clinically significant history of skin disorder (eczema, psoriasis, etc.), allergy, immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness, psychiatric disorder, drug or alcohol abuse.
* Oral or systemic steroid medication or the use of immunosuppressive agents.
* Positive HIV antibody test, HCV antibody test or positive HBV serology except post-vaccination.
* Heaf test greater than Grade II
* Confirmed pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2004-02; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
The occurence and severity of local side-effects The occurence and severity of systemic side-effects | 1 year

SECONDARY OUTCOMES:
The induction of T cell responses (as measured by an interferon-gamma Elispot assay). Other exploratory cellular immunology assays will be performed as such assays are developed. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] McShane H, Brookes R, Gilbert SC, Hill AV. Enhanced immunogenicity of CD4(+) t-cell responses and protective efficacy of a DNA-modified vaccinia virus Ankara prime-boost vaccination regimen for murine tuberculosis. Infect Immun. 2001 Feb;69(2):681-6. doi: 10.1128/IAI.69.2.681-686.2001. PMID 11159955
- [Background] McShane H, Behboudi S, Goonetilleke N, Brookes R, Hill AV. Protective immunity against Mycobacterium tuberculosis induced by dendritic cells pulsed with both CD8(+)- and CD4(+)-T-cell epitopes from antigen 85A. Infect Immun. 2002 Mar;70(3):1623-6. doi: 10.1128/IAI.70.3.1623-1626.2002. PMID 11854254
- [Derived] Whelan KT, Pathan AA, Sander CR, Fletcher HA, Poulton I, Alder NC, Hill AV, McShane H. Safety and immunogenicity of boosting BCG vaccinated subjects with BCG: comparison with boosting with a new TB vaccine, MVA85A. PLoS One. 2009 Jun 16;4(6):e5934. doi: 10.1371/journal.pone.0005934. PMID 19529780